CLINICAL TRIAL: NCT07010822
Title: A Phase III, Double-blind, Randomized, Placebo Controlled Study to Evaluate the Mucosal Intestinal Immunity to Poliovirus Type-2 of nOPV2 at Birth Dose in Healthy IPV Vaccinated Infants
Brief Title: A Study to Evaluate the Mucosal Intestinal Immunity to Poliovirus Type-2 of nOPV2 at Birth Dose in Healthy IPV Vaccinated Infants
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fidec Corporation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: nOPV2-003; INV-081593 (Other Grant/Funding Number: Gates Foundation)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Poliomyelitis
Keywords: Polio; nOPV2; immunity
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- nOPV2 at birth (Experimental): Approximately 330 subjects to receive 1 dose of nOPV2 at birth followed by a regular IPV schedule at approx. 6, 10, 14 weeks of age and an nOPV2-002 challenge at approx. 18 weeks of age.
  Interventions: Biological: nOPV2
- nOPV2 at birth and Wk 14 of age (Experimental): Approximately 80 subjects to receive 2 doses of nOPV2 at birth and 14 wks of age plus a regular IPV schedule at approx. 6, 10, 14 weeks of age and an nOPV2-002 challenge at approx. 18 weeks of age.
  Interventions: Biological: nOPV2
- Placebo (Placebo Comparator): Approximately 330 subjects to receive 2 doses of placebo at birth and 14 wks of age plus a regular IPV schedule at approx. 6, 10, 14 weeks of age and an nOPV2-002 challenge at approx. 18 weeks of age
  Interventions: Biological: nOPV2

INTERVENTIONS:
Biological: nOPV2 — nOPV2 will be administered at birth and Wk 14 of age depending on the study arm.

SUMMARY:
The study will compare the transmissible levels of poliovirus type-2 detected in stool samples collected at the time of the nOPV2 challenge and subsequent timepoints in 3 groups of newborns receiving an nOPV2 dose at birth and primed with 3 doses of IPV (6 - 10 - 14 weeks of age).

DETAILED DESCRIPTION:
To meet the urgent public health need regarding cVDPV2 outbreaks, a novel type 2 OPV (nOPV2) vaccine was developed using attenuated serotype 2 polioviruses derived from a modified Sabin 2 infectious cDNA clone generated by modifying the Sabin-2 ribonucleic acid (RNA) sequence to improve genetic stability and make the strains less prone to reversion to virulence. Clinical trials in adults, children, and infants demonstrated that nOPV2 vaccine is safe, well tolerated, and immunogenic. These include a phase 2 study of vaccine-naïve neonates in Bangladesh who received either two doses of nOPV2 or two doses of placebo at birth and 4 weeks of age concluded that the vaccine was well tolerated and immunogenic, as 90% of the infants seroconverted at 2 weeks post second dose. Overall 99% of infants had protective levels of neutralizing antibody at this time in contrast to the seroprotection rate of 56% in the placebo group.

Although immunogenic, the effect of nOPV2 on virus transmission is still unclear. This phase 3 study aims to compare the transmissible levels of poliovirus type-2 detected in stool samples collected at the time of the nOPV2 challenge (pre-challenge) and subsequent timepoints in 3 groups of newborns receiving an nOPV2 dose at birth and primed with 3 doses of IPV (6 - 10 - 14 weeks of age).

ELIGIBILITY:
Inclusion Criteria:

1. Newborn infants of maximum 1 week of age with birth weight > 2,500 g.
2. Healthy infants without obvious medical conditions like immunodeficiency diseases, severe congenital malformations, severe neurological diseases or any other disease that require high doses of corticosteroids or immunotherapies that preclude the subject from participating in the study as established by medical history and physical examination.
3. Written informed consent obtained from both parents or legal guardian(s) as per country regulations.
4. Resides in the area and parents willing to adhere to all study procedures.

Exclusion Criteria:

1. Any confirmed or suspected immunosuppressive or known immunodeficient condition including human immunodeficiency virus infection in the potential participant or any member of the participant's household.
2. Household member who has receive any novel OPV 1 month before birth of this study's participant up through 1 month post-last-dose.
3. Family history of congenital or hereditary immunodeficiency.
4. Major congenital defects or serious uncontrolled chronic illness (neurologic, pulmonary, gastrointestinal, hepatic, renal, or endocrine).
5. Known allergy to any component of the study vaccines or to any antibiotics that share molecular composition with a component of the study vaccines.
6. Uncontrolled coagulopathy or blood disorder contraindicating intramuscular injections (of IPV)
7. Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
8. Acute severe febrile illness (≥37.5 °C) on the day of vaccination deemed by the Investigator to be a contraindication for vaccination (the child can be included at a later time if within age window and all inclusion criteria are met.).
9. Participant who, in the opinion of the Investigator, is unlikely to comply with the protocol or is inappropriate to be included in the study for the safety or the benefit-risk ratio of the participant.
10. Infants from multiple births or born prematurely (< 37 weeks of gestation).

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 740 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2026-09-21 (Estimated); Study Completion 2026-09-21 (Estimated)

PRIMARY OUTCOMES:
Stool viral load | From enrollment to the end of the study at Wk 22 of age.
  To assess the presence or absence of "transmissible" levels of virus in stool, with presence defined as a log10 CCID50 per gram of ≥4.3 at Visit 7 (Day 126; day of nOPV2 challenge dose administration), Visit 8 (Day 130), Visit 9 (Day 133), Visit 10 (Day 140), and Visit 11 (Day 154) in all groups.

SECONDARY OUTCOMES:
PV Type 2 neutralizing activity in stool samples | From enrollment to the end of the study at 22 Wks of age.
  To assess poliovirus type-2-specific neutralizing activity and total concentrations and poliovirus type-2-specific IgA/IgG mean fluorescence intensities (MFI) in stool samples at Visit 7 (Day 126), Visit 8 (Day 130), Visit 9 (Day 133), Visit 10 (Day 140), and Visit 11 (Day 154) in all groups.
PV Type 2 seroprotection rate | From enrollment till 18 Wks of age
  To assess the seroprotection (SP) rate to poliovirus type-2 on Day 42 (Visit 4) and Week 18 (Visit 7). SP rate is defined as the percentage of subjects with type 2-specific antibody titers ≥ 1:8 in all groups.
PV Type 2 seroconversion rate | From enrollment till Wk 18 of age.
  To assess the seroconversion (SC) rate of poliovirus type-2 neutralizing antibodies on Week 18 (Visit 7) of age in all groups.
PV Type 2 neutralization titers | From enrollment till Wk 18 of age
  To assess the geometric mean and median poliovirus type-2-specific neutralization titers on Week 6 (Visit 4) and Week 18 (Visit 7) of age in all groups.
SAEs and IMEs | From enrollment to the end of the study at Wk 22 of age
  Incidence of SAEs and IMEs by severity and by causal association from the date of informed consent throughout the study period in all groups.
Solicited AEs | From enrollment to Wk 18 of age
  Incidence of mild, moderate and severe solicited AEs (fever, vomiting, abnormal crying, drowsiness, loss of appetite, diarrhea and irritability) for 7 days after each dose of study vaccine/placebo in all groups.
Viral shedding | From enrollment to the end of the study at Wk 22 of age.
  To assess the positivity rate in the poliovirus type-specific RT-PCR assay at Visit 7 (Day 126; day of nOPV2 challenge dose administration), Visit 8 (Day 130), Visit 9 (Day 133), Visit 10 (Day 140), and Visit 11 (Day 154) in all groups.

CONTACTS AND LOCATIONS:
Overall Officials: Khaelqu Zaman, Dr., Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- icddr,b - Matlab Health Research Centre, Chāndpur, Dhaka Division, Bangladesh

IPD SHARING:
Plan to Share IPD: No